CLINICAL TRIAL: NCT06872554
Title: Effects of a Pre Surgery Multicomponent Training Program on Strength, Pain, and Quality of Life in Patients with Abdominal Wall Hernias
Brief Title: Effects of a Multicomponent Training Program on Health Outcomes in Patients with Abdominal Wall Hernia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: University Hospital Virgen del Rocio, Sevilla (Unknown)
Responsible Party: Principal Investigator, Borja Sañudo, Head of the Department of Physical Education and Sport, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID2022-142316OB-I02
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Wall Hernia; Prevention; Exercise; Physical Activity
Keywords: hernia; abdominal wall; exercise intervention; quality of life; pain; incisional hernial
MeSH Terms: conditions — Hernia, Abdominal; Motor Activity; Hernia; Pain

STUDY DESIGN:
Intervention Model Description: The following study is a randomized clinical trial consisting of three parallel arms. Stratified randomization will be performed to allocate subjects into the three groups (supervised intervention, unsupervised intervention, and control group). Subjects with 12 weeks or less until surgery will be randomized between the supervised intervention group and the control group. Subjects with more than 12 weeks until surgery will be included in the unsupervised intervention group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Supervised Exercise Intervention (Experimental): Group that will follow the 12-week training program supervised by a professional in physical activity and sports sciences.
  Interventions: Other: Supervised exercise training
- Non Supervised Exercise Intervention (Active Comparator): Group that will follow the 12-week training program from home, without the supervision of a professional in physical activity and sports sciences.
  Interventions: Other: Non supervised exercise training
- Control Group (No Intervention): Participants randomly assigned to the control group will receive advice on the importance of an active lifestyle for their quality of life.

INTERVENTIONS:
Other: Supervised exercise training — The intervention will consist of a 12-week multicomponent training program. This program will include exercises focused on strength training, mobility, stretching, and breathing. Throughout the 12 weeks, there will be a progressive increase in training volume-understood as the number of sets and repetitions performed-and in intensity, defined as the difficulty involved in performing the exercises. After each training session, data will be collected on the perceived effort and the pain in the area affected by the abdominal hernia.
  Arms: Supervised Exercise Intervention
Other: Non supervised exercise training — The intervention will consist of a 12-week multicomponent training program. This program will include exercises focused on strength training, mobility, stretching, and breathing. Throughout the 12 weeks, there will be a progressive increase in training volume-understood as the number of sets and repetitions performed-and in intensity, defined as the difficulty involved in performing the exercises. After each training session, data will be collected on the perceived effort and the pain in the area affected by the abdominal hernia. This program will be realized for the participants at home, with the use of a specified training App, without the supervision of a sport science professional.
  Arms: Non Supervised Exercise Intervention

SUMMARY:
Abdominal wall hernias are among the most prevalent pathologies today, characterized by specific symptoms such as pain, a sensation of tightness in the affected area, and potential gastrointestinal complications. These symptoms negatively impact patients' health and quality of life.

In other clinical conditions, such as osteoarthritis, sarcopenia, and fibromyalgia, participation in multicomponent training programs (which integrate strength, mobility, and stretching exercises) has been documented to significantly improve quality of life, reduce pain, and optimize patients' functional capacity. Likewise, scientific literature highlights that in the context of injuries requiring surgical intervention, such as anterior cruciate ligament or meniscus tears, patients who underwent prehabilitation programs based on multicomponent training experienced fewer losses in functional and structural aspects, such as strength and muscle mass. These programs also contributed to a reduction in postoperative pain perception.

Therefore, the primary objective of this study is to evaluate the effects of a multicomponent training program on health variables (pain, quality of life, perceived exertion, and recurrence) and functional capacity (trunk isometric strength, grip strength, and lower limb dynamic strength) in patients with abdominal wall hernias. As a secondary objective, the impact of this program on the aforementioned variables after abdominal wall repair surgery will be investigated.

DETAILED DESCRIPTION:
Background:

Abdominal wall hernias are one of the most prevalent pathologies in contemporary clinical practice, affecting a significant percentage of the global population. These hernias, characterized by the protrusion of organs or tissues through a weakened area in the abdominal musculature, may present symptoms such as pain, tightness, and gastrointestinal complications, impacting both general health and patients' quality of life. The management of these conditions often involves surgical intervention, with variable outcomes in terms of functional recovery and postoperative pain. However, there are still opportunities to improve preoperative and postoperative treatment strategies through comprehensive approaches that include adapted physical training programs.

In recent years, the field of physical rehabilitation has advanced significantly due to the development of multicomponent training programs. These programs, combining strength, mobility, and stretching exercises, have proven effective in improving quality of life and reducing pain in various chronic pathologies. For instance, in patients with osteoarthritis, multicomponent training has been shown not only to mitigate pain but also to improve functional capacity and reduce progressive joint deterioration. In sarcopenia, a common problem in older adults, resistance training has demonstrated significant benefits in maintaining muscle mass and strength, contributing to a better quality of life.

Moreover, participation in prehabilitation programs has been particularly beneficial in the context of surgical procedures. Recent studies have documented that patients undergoing anterior cruciate ligament or meniscal interventions who participated in multicomponent prehabilitation programs experienced less strength and muscle mass loss, as well as a reduced perception of postoperative pain. A recent meta-analysis also shows that prehabilitation programs including strength training and aerobic exercises contributed to improved functional outcomes and shorter hospital stays in patients undergoing major abdominal surgery. This proactive approach, which prepares the body for surgical stress, has proven to be an effective strategy for improving postoperative outcomes and accelerating recovery.

However, despite evidence supporting the use of multicomponent training programs in other clinical and surgical conditions, their application in patients with abdominal wall hernias has been scarcely explored. The current literature lacks studies that comprehensively address the impact of prehabilitation in this patient group, both in the preoperative phase and postoperative recovery. Given that hernia repair surgery is one of the most common surgical interventions, with significant implications for functional capacity and overall well-being, implementing prehabilitation strategies based on multicomponent training could represent an important innovation in managing these conditions.

In conclusion, this study proposes that a multicomponent prehabilitation program could not only improve functional capacity and reduce preoperative pain in patients with abdominal wall hernias but also optimize postoperative outcomes and overall recovery. This approach is based on accumulated evidence in other clinical and surgical fields, reinforcing the need to explore its applicability and effectiveness in this specific context.

Study Objectives:

Evaluate the effects of a multicomponent training program on strength levels, quality of life, and pain in patients with abdominal wall hernias.

Assess the effects of the multicomponent training program on the aforementioned variables post-abdominal wall surgery.

Determine how the intervention affects hospital stay duration and postoperative complications.

Analyze differences between supervised and unsupervised training programs.

Compare postoperative functional recovery between the intervention and control groups.

Methodology:

An experimental, prospective, and longitudinal study will be conducted, implementing a multicomponent training program over 12 weeks. Patients will be recruited from the Abdominal Wall Surgery Unit of Virgen del Rocío Hospital.

Inclusión Criteria:

Patients ≥ 18 years; Ventral hernia ≥ 4cm (W2-3 per EHS classification); Signed informed consent.

Exclusión Criteria:

Patients <18 years; Ventral hernia <4cm (W1 per EHS classification); Severe physical/cognitive impairment affecting mobility and daily activities.

Study Phases:

1. Patient Recruitment: Eligible patients will be randomized into three groups: supervised intervention, online intervention, and control.
2. Data Collection: Muscle strength, pain, quality of life, perceived exertion, and body composition will be evaluated pre-intervention, post-intervention, and three months post-surgery.
3. Statistical Analysis: Descriptive and multivariate statistical models will be applied to determine associations between intervention and study variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Ventral hernia ≥ 4cm (W2-3 per EHS classification)
* Signed informed consent

Exclusion Criteria:

* Patients <18 years
* Ventral hernia <4cm (W1 per EHS classification)
* Severe physical/cognitive impairment affecting mobility and daily activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Abdominal Muscles Wall Strength | Pre (0 week), Post (12 week), Post Surgery (3 month)
  To assess the strength of the abdominal wall muscles, the isometric trunk flexion test in a seated position will be used, both in the sagittal and transverse planes, utilizing a strain gauge (Chronojump, Barcelona, Spain). The variables collected will be the maximum isometric strength and the rate of force development.
Health Releated Quality of Life | Pre (0 week), Post (12 week), Post Surgery (1 month), Post Surgery (3 month)
  Quality of life will be assessed using a specific questionnaire for abdominal wall hernias (HerQLes) and a general questionnaire (SF 12)
Pain | Pre (0 week), Post (12 week), Post Surgery (1 month), Post Surgery (3 month)
  Pain will be assessed using a visual analog scale (VAS), where 0 represents no pain and 10 represents maximum pain.

SECONDARY OUTCOMES:
Physical Activity Level | Pre (0 week)
  The level of physical activity will be assessed using the IPAQ Short Version questionnaire, which assess the physical activity on the las 7 days.
Sedentary Behaviour | Pre (0 week)
  The level of sedentary behavior will be assessed using the Sedentary Behavior Questionnaire (SBQ), which evaluates the time a person spends sitting on weekdays and weekends.
Physical Performance | Pre (0 week), Post (12 week), Post Surgery (3 month)
  To assess physical abilities, three tests from the Senior Fitness Test will be used: handgrip strength, sit-to-stand in 30 seconds, and walking speed over 4 meters.
Body Composition | Pre (0 week), Post (12 week), Post Surgery (3 month)
  Muscle mass, fat mass, weight, and body mass index (BMI) will be evaluated using a digital bioimpedance scale (TANITA BC 545N).

CONTACTS AND LOCATIONS:
Overall Officials: Borja Sañudo Corrales, Phd, Study Director — University of Seville

IPD SHARING:
Plan to Share IPD: Undecided
Once processing, quality control, analysis and publication are complete, the data will be made accessible in open access repositories. These data will be anonymized (remove potentially identifying information).